CLINICAL TRIAL: NCT00617890
Title: A Study to Determine the Activity of SCH 717454 in Subjects With Osteosarcoma or Ewing's Sarcoma That Has Relapsed After Standard Systemic Therapy
Brief Title: A Study to Determine the Activity of Robatumumab (SCH 717454) in Participants With Relapsed Osteosarcoma or Ewing's Sarcoma (MK-7454-002/P04720)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated for strategic reasons, not for a safety concern.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04720
Record Dates: First submitted 2008-01-17; First posted 2008-02-18 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Osteosarcoma; Sarcoma, Ewing's; Peripheral Neuroectodermal Tumor
Keywords: anti-IGF-1R
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral | interventions — robatumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: 0.3 mg/kg (Experimental): Participants received robatumumab 0.3 mg/kg intravenously (IV) as a single dose on Day 1, followed by surgery on Day 10 to 14, and four weeks later, resumption of robatumumab 0.3 mg/kg on the same calendar day (± 3 days) once every 2 weeks until disease recurrence or up to 1 year of dosing. This group comprised participants with resectable osteosarcoma that relapsed within 6 months of prior definitive treatment (eg surgical metastasectomy) and having at least one prior chemotherapy regimen containing a platinum agent and doxorubicin.
  Interventions: Biological: robatumumab
- Group 1: 10 mg/kg (Experimental): Participants who received robatumumab 10 mg/kg IV as a single dose on Day 1, followed by surgery on Day 10 to 14, and four weeks later, resumption of robatumumab 10 mg/kg on the same calendar day (± 3 days) once every 2 weeks until disease recurrence or up to 1 year of dosing. This group comprised participants with resectable osteosarcoma that relapsed within 6 months of prior definitive treatment (eg surgical metastasectomy) and having at least one prior chemotherapy regimen containing a platinum agent and doxorubicin.
  Interventions: Biological: robatumumab
- Group 2: 10 mg/kg (Experimental): Participants received robatumumab 10 mg/kg IV biweekly until disease recurrence or up to 1 year of dosing. This group comprised participants with relapsed and unresectable osteosarcoma refractory to prior chemotherapy with a platinum- and doxorubicin-containing regimen.
  Interventions: Biological: robatumumab
- Group 3: 10 mg/kg (Experimental): Participants received robatumumab 10 mg/kg IV biweekly until disease recurrence or up to 1 year of dosing. This group comprised participants with Ewing sarcoma refractory to prior treatment with at least 3 of the following agents: ifosfamide, etoposide, cyclophosphamide, doxorubicin, or vincristine.
  Interventions: Biological: robatumumab

INTERVENTIONS:
Biological: robatumumab — Robatumumab IV every two weeks until disease progression.
  Other Names: SCH 717454; SCH 717454 (19D12); MK-7454

SUMMARY:
Participants with relapsed osteosarcoma that can be treated with surgery will be randomized to robatumumab administered intravenously (IV) at one of two dose levels. These participants will first receive robatumumab, have surgery performed, and continue to receive treatment every two weeks until a year of dosing, or until disease progression.

Participants with unresectable osteosarcoma or Ewing Sarcoma will receive robatumumab IV once every two weeks until disease progression. Participants who achieve a complete response (CR) or partial response (PR) after tumor evaluations may undergo surgical resection. After surgery, participants are eligible to receive 10 mg/kg robatumumab until disease recurrence/progression or one year of total dosing, whichever occurs first.

DETAILED DESCRIPTION:
Participants with resectable osteosarcoma will be randomized to one of two dose levels of robatumumab to be given intravenously. These participants will first receive robatumumab according to randomized treatment, and have surgery performed 10 to 14 days after initial dosing. Participants will be allowed to recover from surgery four to six weeks prior to additional robatumumab administration at their randomized dose level. robatumumab will then be administered on the same calendar day once every two weeks. Participants will continue to receive robatumumab until disease recurrence, or until completing a year of dosing at the same dose level assigned, whichever occurs first.

Participants with unresectable osteosarcoma or Ewing Sarcoma will be assigned treatment to robatumumab IV administered once every two weeks and will continue to receive robatumumab until disease progression. Participants who achieve a CR or PR after tumor evaluations may undergo surgical resection. After surgery, participants are eligible to receive 10 mg/kg robatumumab until disease recurrence/progression or one year of total dosing, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* A participant must be 11 years of age or older and may be of any race, and gender; participants between 4 and 10 years of age, inclusive, may be considered on a site-by-site basis.
* A participant must have a diagnosis of histologically confirmed osteosarcoma or Ewing sarcoma;
* A participant with either:

  * relapsed and resectable osteosarcoma
  * relapsed and unresectable osteosarcoma that is refractory to standard therapy, ie. has relapsed after prior systemic treatment with active chemotherapy agents
  * Ewing sarcoma that is refractory to standard systemic therapies
* A participant >16 years of age must have an Eastern Cooperative Oncology Group (ECOG) performance status of <=2; a participant <=16 years of age must have a Karnofsky performance status between 50% and 100% or a Lansky play scale between 50% and 100%
* A participant must have adequate organ function.

Exclusion Criteria:

* A participant with a history of another malignancy (with the exception of non-melanoma skin cancer or carcinoma in situ of the cervix treated with curative intent at least 2 years prior to start of treatment, or other adequately treated malignancy for which the subject has been disease free for >=5 years)
* A participant who has known treated or untreated leptomeningeal metastasis, or a metastatic central nervous system lesion
* A participant with a history of uncontrolled diabetes mellitus
* A participant with a recent myocardial infarction (within the past year); or a participant who at the time of Screening presents with unstable or uncontrolled angina, New York Heart Association (NYHA) Class III or IV congestive heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram (ECG) abnormality
* A participant with an active infection
* A participant with clinically significant hepatitis at Screening, or a participant who is hepatitis C antibody positive, hepatitis B surface antigen positive, or human immunodeficiency virus (HIV) seropositive
* A participant who has been treated with an anti-insulin-like growth factor receptor 1 (anti-IGF-1R)- targeted drug or antibody
* A participant with known hypersensitivity to other antibodies, or any accompanying excipients associated with these medications.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2011-08-31 (Actual); Study Completion 2013-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Anderson PM, Bielack SS, Gorlick RG, Skubitz K, Daw NC, Herzog CE, Monge OR, Lassaletta A, Boldrini E, Papai Z, Rubino J, Pathiraja K, Hille DA, Ayers M, Yao SL, Nebozhyn M, Lu B, Mauro D. A phase II study of clinical activity of SCH 717454 (robatumumab) in patients with relapsed osteosarcoma and Ewing sarcoma. Pediatr Blood Cancer. 2016 Oct;63(10):1761-70. doi: 10.1002/pbc.26087. Epub 2016 Jun 30. PMID 27362300
- [Derived] Asmane I, Watkin E, Alberti L, Duc A, Marec-Berard P, Ray-Coquard I, Cassier P, Decouvelaere AV, Ranchere D, Kurtz JE, Bergerat JP, Blay JY. Insulin-like growth factor type 1 receptor (IGF-1R) exclusive nuclear staining: a predictive biomarker for IGF-1R monoclonal antibody (Ab) therapy in sarcomas. Eur J Cancer. 2012 Nov;48(16):3027-35. doi: 10.1016/j.ejca.2012.05.009. Epub 2012 Jun 7. PMID 22682017
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04720&kw=P04720&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 10 mg/kg: Participants received robatumumab 10 mg/kg IV as a single dose on Day 1, followed by surgery on Day 10 to 14, and four weeks later, resumption of robatumumab 10 mg/kg on the same calendar day (± 3 days) once every 2 weeks until disease recurrence or up to 1 year of dosing. This group comprised participants with resectable osteosarcoma that relapsed within 6 months of prior definitive treatment (eg surgical metastasectomy) and having at least one prior chemotherapy regimen containing a platinum agent and doxorubicin.
- Group 3: 10 mg/kg: Participants received robatumumab 10 mg/kg IV biweekly until disease recurrence or up to 1 year of dosing. This group comprised participants with Ewing's sarcoma refractory to prior treatment with at least 3 of the following agents: ifosfamide, etoposide, cyclophosphamide, doxorubicin, or vincristine.
Period: Overall Study
Arm/Group | Group 1: 0.3 mg/kg | Group 1: 10 mg/kg | Group 2: 10 mg/kg | Group 3: 10 mg/kg
Started | 35 | 33 | 35 | 116
Received Treatment | 34 | 33 | 34 | 115
Completed | 4 | 5 | 0 | 1
Not Completed | 31 | 28 | 35 | 115
Not completed — Treatment ongoing at data cut-off | 0 | 0 | 0 | 5
Not completed — Lack of Efficacy | 23 | 26 | 30 | 97
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 2
Not completed — Protocol Violation | 2 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 3 | 8
Not completed — Not treated | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Three participants did not receive study treatment but are included in the baseline population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 0.3 mg/kg | Group 1: 10 mg/kg | Group 2: 10 mg/kg | Group 3: 10 mg/kg | Total
Number analyzed (Participants) | 35 | 33 | 35 | 116 | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.7 (15.5) | 20.1 (10.3) | 27.5 (15.3) | 24.6 (11.4) | 24.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 11 | 43 | 81
  Male | 21 | 20 | 24 | 73 | 138

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Complete Response or Partial Response (Group 3 Only)
Description: This is a measure of the number of participants with a complete response (CR) or partial response (PR) to therapy, confirmed by central review. Response was based on Response Evaluation Criteria in Solid Tumors (RECIST) and World Health Organization (WHO) criteria.
Time Frame: Up to 1 year following the start of study therapy
Population: Participants in Group 3 with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Group 3: 10 mg/kg
Number analyzed (Participants) | 84
Participants | 6

2. Primary Outcome: Number of Participants With >= 25% Change in Tumor Proliferation After Exposure to Robatumumab (Group 1 Only)
Description: Tumor proliferation was measured using Ki-67 levels. Ki-67 is nuclear protein associated with cellular proliferation.
Time Frame: Approximately 14 days
Population: Group 1 Participants; this outcome was not evaluated due to early termination of the study.
Arm/Group | Group 1: 0.3 mg/kg | Group 1: 10 mg/kg
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Participants Achieving a Complete Response, a Partial Response, or Stable Disease (Group 2 Only)
Description: Responses to treatment (complete response, partial response, or stable disease) confirmed by central review for Participants in Group 2. Response was based on Response Evaluation Criteria in Solid Tumors (RECIST) and World Health Organization (WHO) criteria.
Time Frame: Up to 1 year following the start of study therapy
Population: Group 2 participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Group 2: 10 mg/kg
Number analyzed (Participants) | 29
Participants | 6

4. Secondary Outcome: Overall Survival
Description: This is a measure of the number of participants known to be alive at the time of data analysis for this study.
Time Frame: From start of treatment until death or data analysis cut off (Up to 3.4 years)
Population: All study participants
Measure: Number; unit: Participants
Arm/Group | Group 1: 0.3 mg/kg | Group 1: 10 mg/kg | Group 2: 10 mg/kg | Group 3: 10 mg/kg
Number analyzed (Participants) | 35 | 33 | 35 | 116
Participants | 17 | 16 | 7 | 28

5. Secondary Outcome: Time Until Tumor Relapse (Group 1 Only)
Description: This is a measure of the time from the start of the study to documented relapse of disease.
Time Frame: From start of treatment until relapse or data analysis cut off (Up to 3.4 years)
Population: Group 1 participants; this outcome was not evaluated due to early termination of the study.
Arm/Group | Group 1: 0.3 mg/kg | Group 1: 10 mg/kg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of Serum Levels of Robatumumab (Group 1 Only)
Time Frame: End of infusion on Day 1, and then prior to surgery, before and after the 2nd, 3rd, and 8th doses (up to 20 weeks)
Population: Group 1, both dose levels: this outcome was not evaluated due to early termination of the study.
Arm/Group | Group 1: 0.3 mg/kg | Group 1: 10 mg/kg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Anti-robatumumab Antibodies
Description: For biological agents, it is possible for the host (participant) to develop antibodies to the agent. This outcome measure was planned to find out the number of participants who developed the antibodies after treatment with robatumumab.
Time Frame: Up to 2 years
Population: This outcome was not evaluated due to early termination of the study.
Arm/Group | Group 1: 0.3 mg/kg | Group 1: 10 mg/kg | Group 2: 10 mg/kg | Group 3: 10 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment. Treatment-emergent adverse events are those that occur after participants have received study treatment, or existing adverse events that occurred during screening that increase in severity after study treatment. Adverse events in the Group 1: 0.3 mg/kg arm that occurred after switching to the 10 mg/kg dose are displayed under the originally assigned treatment.
Time Frame: Up to 2 years
Population: All participants receiving study drug.
Measure: Number; unit: Participants
Arm/Group | Group 1: 0.3 mg/kg | Group 1: 10 mg/kg | Group 2: 10 mg/kg | Group 3: 10 mg/kg
Number analyzed (Participants) | 34 | 33 | 34 | 115
Participants | 31 | 30 | 31 | 112

9. Secondary Outcome: Time to Disease Progression (Groups 2 and 3 Only)
Description: This is a measure of the time from the start of the study to the time of documented disease progression.
Time Frame: From the start of treatment until disease progression or data analysis cut off (Up to 3.4 years)
Population: All participants in Groups 2 and 3; this outcome was not evaluated due to early termination of the study
Arm/Group | Group 2: 10 mg/kg | Group 3: 10 mg/kg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Overall Survival (Groups 2 and 3 Only)
Description: This is a measure of the time of survival from first dose to documentation of death
Time Frame: From start of treatment until death or data analysis cut off (Up to 3.4 years)
Population: Group 2 and 3 Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 2: 10 mg/kg | Group 3: 10 mg/kg
Number analyzed (Participants) | 35 | 116
Months | 8.18 [2.96 to 10.58] | 6.93 [4.93 to 11.10]

11. Secondary Outcome: Duration of Response (Groups 2 and 3 Only)
Description: This is a measure of the amount of time in which the tumor responded to therapy.
Time Frame: From time of documented response until disease progression or data analysis cut off (Up to 3.4 years)
Population: Group 2 and 3 participants; this outcome was not evaluated due to early termination of the study
Arm/Group | Group 2: 10 mg/kg | Group 3: 10 mg/kg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are reported from enrollment up to 5 weeks after the end of treatment (up to 2 years)
Description: All treated participants; adverse events in the Group 1: 0.3 mg/kg arm that occurred after switching to the 10 mg/kg dose are displayed under the originally assigned treatment.
Groups:
- Group 1: 0.3mg/kg: Participants received robatumumab 0.3 mg/kg intravenously (IV) as a single dose on Day 1, followed by surgery on Day 10 to 14, and four weeks later, resumption of robatumumab 0.3 mg/kg on the same calendar day (± 3 days) once every 2 weeks until disease recurrence or up to 1 year of dosing. This group comprised participants with resectable osteosarcoma that relapsed within 6 months of prior definitive treatment (eg surgical metastasectomy) and having at least one prior chemotherapy regimen containing a platinum agent and doxorubicin.
- Group 1: 10mg/kg: Participants received robatumumab 10 mg/kg IV as a single dose on Day 1, followed by surgery on Day 10 to 14, and four weeks later, resumption of robatumumab 10 mg/kg on the same calendar day (± 3 days) once every 2 weeks until disease recurrence or up to 1 year of dosing. This group comprised participants with resectable osteosarcoma that relapsed within 6 months of prior definitive treatment (eg surgical metastasectomy) and having at least one prior chemotherapy regimen containing a platinum agent and doxorubicin.
- Group 2: 10mg/kg: Participants received robatumumab 10 mg/kg IV biweekly until disease recurrence or up to 1 year of dosing. This group comprised participants with relapsed and unresectable osteosarcoma refractory to prior chemotherapy with a platinum- and doxorubicin-containing regimen.
- Group 3: 10mg/kg: Participants received robatumumab 10 mg/kg IV biweekly until disease recurrence or up to 1 year of dosing. This group comprised participants with Ewing's sarcoma refractory to prior treatment with at least 3 of the following agents: ifosfamide, etoposide, cyclophosphamide, doxorubicin, or vincristine.
Arm/Group | Group 1: 0.3mg/kg | Group 1: 10mg/kg | Group 2: 10mg/kg | Group 3: 10mg/kg
Serious Adverse Events (participants affected / at risk) | 17/34 | 8/33 | 12/34 | 57/115
Other Adverse Events (participants affected / at risk) | 28/34 | 30/33 | 29/34 | 104/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 0.3mg/kg (N=34) | Group 1: 10mg/kg (N=33) | Group 2: 10mg/kg (N=34) | Group 3: 10mg/kg (N=115)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (6)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APLASIA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
BLINDNESS UNILATERAL (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
CONDITION AGGRAVATED (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEVICE DISLOCATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTHERMIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 11 (13)
PERFORMANCE STATUS DECREASED (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (11)
HEPATIC HAEMORRHAGE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CENTRAL NERVOUS SYSTEM INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
BRAIN HERNIATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE RESPIRATORY DISTRESS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WOUND NECROSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BIOPSY BONE ABNORMAL (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERCREATINAEMIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOSARCOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COMA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENINGEAL DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOCLONUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NERVE COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BRONCHIAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY TOXICITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 5 (5)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEG AMPUTATION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MEDICAL DEVICE REMOVAL (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THORACOTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WOUND TREATMENT (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 0.3mg/kg (N=34) | Group 1: 10mg/kg (N=33) | Group 2: 10mg/kg (N=34) | Group 3: 10mg/kg (N=115)
ANAEMIA (Blood and lymphatic system disorders) | 6 (8) | 2 (3) | 3 (4) | 22 (44)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 17 (35)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
TINNITUS (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 9 (13)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 9 (10)
CONSTIPATION (Gastrointestinal disorders) | 9 (9) | 9 (10) | 3 (3) | 34 (43)
DIARRHOEA (Gastrointestinal disorders) | 3 (6) | 6 (11) | 2 (2) | 29 (42)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2) | 4 (5)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
NAUSEA (Gastrointestinal disorders) | 13 (20) | 12 (18) | 5 (6) | 35 (48)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 6 (6)
VOMITING (Gastrointestinal disorders) | 9 (12) | 8 (9) | 3 (4) | 25 (40)
ASTHENIA (General disorders) | 0 (0) | 1 (4) | 1 (1) | 13 (18)
CHEST PAIN (General disorders) | 7 (8) | 3 (3) | 3 (3) | 10 (12)
FATIGUE (General disorders) | 7 (10) | 7 (8) | 7 (7) | 23 (28)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 2 (7) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 2 (2) | 3 (3) | 4 (4)
PAIN (General disorders) | 4 (4) | 4 (4) | 2 (2) | 9 (11)
PYREXIA (General disorders) | 9 (11) | 11 (13) | 6 (7) | 21 (37)
BRONCHITIS (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (2)
RHINITIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
SINUSITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 5 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (7) | 3 (4) | 1 (1) | 7 (13)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 8 (12)
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
POST-THORACOTOMY PAIN SYNDROME (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 13 (16) | 6 (7) | 1 (1) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (11)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 9 (11)
HAEMOGLOBIN DECREASED (Investigations) | 5 (6) | 6 (12) | 1 (1) | 3 (4)
PLATELET COUNT DECREASED (Investigations) | 3 (4) | 1 (1) | 0 (0) | 2 (6)
WEIGHT DECREASED (Investigations) | 1 (1) | 1 (1) | 2 (2) | 11 (13)
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 (6) | 4 (5) | 4 (4) | 27 (37)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 6 (11) | 3 (6) | 1 (1) | 12 (18)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 5 (5)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 2 (2) | 4 (8)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (4) | 2 (3) | 0 (0) | 6 (8)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 1 (1) | 2 (2)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (4) | 3 (3) | 10 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 6 (7) | 15 (19)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 6 (6)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (5)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (6) | 2 (2) | 11 (13)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4) | 7 (8)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 13 (16)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 6 (7)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (8) | 6 (8) | 12 (25)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 8 (11)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (10)
HEADACHE (Nervous system disorders) | 9 (16) | 7 (8) | 7 (10) | 24 (57)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (9)
ANXIETY (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3) | 18 (24)
DEPRESSION (Psychiatric disorders) | 1 (1) | 3 (4) | 2 (2) | 4 (4)
INSOMNIA (Psychiatric disorders) | 4 (4) | 3 (4) | 2 (2) | 20 (20)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (9) | 6 (6) | 16 (19)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4) | 4 (4) | 7 (7)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 2 (2) | 11 (11)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (5) | 0 (0) | 9 (11)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (3) | 2 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 2 (2) | 11 (15)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (2) | 6 (6)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3) | 1 (1) | 2 (2)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (10) | 1 (1) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (6) | 2 (2) | 5 (6)
RASH (Skin and subcutaneous tissue disorders) | 3 (6) | 2 (2) | 1 (1) | 11 (12)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 6 (6)

LIMITATIONS AND CAVEATS:
The study was stopped prematurely for administrative reasons; not all planned endpoints were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the Sponsor. The Investigator further agrees to provide to the Sponsor 45 days prior to submission any publication, presentation, abstracts, manuscripts, or electronic media that report any results of the study. The Sponsor shall have the right to review and comment.